CLINICAL TRIAL: NCT03471377
Title: Improving Planned Surgical Case Duration Accuracy by Leveraging the EHR and Predictive Modeling - A Randomized Control Trial
Brief Title: Improving Planned Surgical Case Duration Accuracy by Leveraging the EHR and Predictive Modeling
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 18-115
Record Dates: First submitted 2018-03-12; First posted 2018-03-20 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Operative Time
Keywords: Planned Surgical Case; Predictive Modeling; 18-115

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- standard scheduling process: Scheduling office assigns start time and room for case and places case on schedule. At this point a default case duration is evaluated by the scheduling office, to see if the value is considered excessively short or excessively long.
  Interventions: Other: standard scheduling process
- assigned a planned case duration value from predictive model: Predictive model calculates new duration for case at 3AM the day before surgery, and the predictions are made available on a SecureShare-site.
  Interventions: Other: assigned a planned case duration value from predictive model

INTERVENTIONS:
Other: standard scheduling process — Scheduling office assigns start time and room for case and places case on schedule. At this point a default case duration is evaluated by the scheduling office, to see if the value is considered excessively short or excessively long. Depending on the assessment, the scheduling office will either keep the default value, use the value that the surgeon placed in the notes (if available), or the scheduling office provides their own estimation.
  Groups: standard scheduling process
Other: assigned a planned case duration value from predictive model — Predictive model calculates new duration for case at 3AM the day before surgery, and the predictions are made available on a SecureShare-site.
  Model predictions are then read by scheduling manager sometime between 7am-10am from the SecureShare site, and the scheduling manager will in EPIC/OpTime, overwrite the current estimate with the new duration value that was generated by the predictive model.
  Groups: assigned a planned case duration value from predictive model

SUMMARY:
The investigators are studying the duration it takes surgeons to complete their respective surgical cases. The hospital hopes to improve the overall operating room scheduling accuracy from this project.

ELIGIBILITY:
Inclusion Criteria:

* A surgeon or OR staff member in the Department of Surgery Gynecology and Colorectal service

Exclusion Criteria:

* Any new surgeon that starts their practice during the study
* Surgery will take place at a location other than the Main hospital or Josie Robertson Surgical Center
* Cases where input data was not available prior to the prediction generation including late add-on cases such as urgent and emergent cases that are placed on the schedule less than 24 hours before the surgery

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Surgeons and OR staff from the GYN and CRS services
Sampling Method: Probability Sample
Enrollment: 683 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
duration it takes surgeons to complete their respective surgical cases | 1 year
  All Gynecology (GYN) and Colorectal (CRS) Surgeons at MSKCC will be included. To test the hypothesis that the developed surgical case duration prediction model compared to the current process of estimating surgical case durations, will show improved prediction accuracy, measured by mean absolute error.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Stromblad, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memoral Sloan Kettering Basking Ridge, New York, New York, United States

REFERENCES:
- [Derived] Stromblad CT, Baxter-King RG, Meisami A, Yee SJ, Levine MR, Ostrovsky A, Stein D, Iasonos A, Weiser MR, Garcia-Aguilar J, Abu-Rustum NR, Wilson RS. Effect of a Predictive Model on Planned Surgical Duration Accuracy, Patient Wait Time, and Use of Presurgical Resources: A Randomized Clinical Trial. JAMA Surg. 2021 Apr 1;156(4):315-321. doi: 10.1001/jamasurg.2020.6361. PMID 33502448
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm